CLINICAL TRIAL: NCT02027220
Title: Phase Ⅱ Study of G-CSF, Bortezomib, Cyclophosphamide and Dexamethasone in Patients With Multiple Myeloma
Brief Title: Combination of G-CSF, Bortezomib, Cyclophosphamide and Dexamethasone in Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, jinxiang fu, M.D., Ph.D., Second Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBCD-001
Record Dates: First submitted 2013-12-21; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Myeloma; Bortezomib; Cyclophosphamide; Dexamethasone; Granulocyte Colony-Stimulating Factor
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Granulocyte Colony-Stimulating Factor; Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- G-CSF/Bortez/Cyc/Dex (Experimental): G-CSF IC on days 0, 1, 7, 8, 14, 15, 21 and 22. Bortezomib IV on days 1, 8, 15 and 22. Cyclophosphamide CIV on days 1, 8, 15 and 22. Dexamethasone IV on days 1, 2, 8, 9, 15, 16, 22 and 23.
  Interventions: Drug: G-CSF; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: G-CSF — G-CSF Intracutaneous injection (IC) on days 0, 1, 7, 8, 14, 15, 21 and 22, every four weeks.
Drug: Bortezomib — Bortezomib Intravenous injection (IV) on days 1, 8, 15 and 22, every four weeks.
  Other Names: Velcade
Drug: Cyclophosphamide — Cyclophosphamide, Continuously Intravenous injection (CIV) on days 1, 8, 15 and 22, every four weeks.
Drug: Dexamethasone — Dexamethasone Intravenous injection (IV) on days 1, 2, 8, 9, 15, 16, 22 and 23, every four weeks.

SUMMARY:
RATIONALE: Bortezomib may stop the growth of myeloma cells by blocking proteasome activity. Cyclophosphamide and dexamethasone may work in different ways to stop the growth of myeloma cells by stopping them from dividing or by killing the cells. Granulocyte Clone Stimulating Factor (G-CSF) possesses the ability to mobilize the plasma cells to detach from myeloma niche, so as to promote drug sensitivity.

PURPOSE: This phase Ⅱ trial is to study how well combination of G-CSF, bortezomib, cyclophosphamide and dexamethasone works in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
Myeloma cells reside in specialised microenvironments, which is called myeloma niche. Myeloma niche provides important cell-cell interactions and signalling molecules that regulate localization and proliferation of myeloma cells. stromal cell-derived factor 1(SDF-1)/Chemokine (C-X-C Motif) Receptor 4 (CXCR4) plays an important role in this process. G-CSF is reported to induce stem cell mobilization by decreasing bone marrow SDF-1. Our in vitro study found that G-CSF enhanced bortezomib activity by inhibiting SDF-1/CXCR4. Myeloma patients treated with Bortezomib, Cyclophosphamide and Dexamethasone have achieved a relatively good response, with an ORR about 80% and complete remission about 40%. We hypothesized that G-CSF may mobilize myeloma cells from myeloma niches thus to enhance bortezomib activity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years, ≤ 80 years.
2. Newly diagnosed multiple myeloma according to International Myeloma Working Group.
3. Relapsed or bortezomib resistant multiple myeloma (MM), who didn't received bortezomib during the last line of therapy for MM prior to this study.
4. Progressive disease according to International Myeloma Working Group.
5. Negative pregnancy test for female with reproductive ability.
6. Signed written informed consent.

Exclusion Criteria:

1. The patient has a history of other active malignancies within 3 years prior to study entry.
2. The patient exhibits evidence of clinically significant uncontrolled conditions including, but not limited to: uncontrolled systemic infection (viral, bacterial, or fungal).
3. Female patient is pregnant or breast-feeding.
4. Known infection with HIV, active Hepatitis B or Hepatitis C.
5. The patient has a history of prior toxicity from bortezomib, cyclophosphamide or dexamethasone that resulted in permanent discontinuation of treatments.
6. Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to study drug administration.
7. Uncontrolled hypertension (defined as systolic blood pressure[BP] > 160 millimeters of mercury (mmHg) or diastolic BP > 100mmHg).
8. Myocardial infarction or unstable angina within the past 6 months prior to study drug administration. Heart failure of New York Heart Association function Class Ⅲ or Ⅳ prior to study drug administration.
9. System illness or other severe concurrent disease or alcoholism, which, in the judgement of the investigator, would make inappropriate for entry into this study or interfere significantly with the proper assessment of safety and efficacy of investigational treatments.
10. Known or suspected of not being able to comply with the trial protocol.
11. Having been previously enrolled in this clinical trial.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 4 months
  Defined as the portion of patients whose best response is equal to or better than partial response (PR), including stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) according to International Myeloma Working Group (IMWG). Response was confirmed after every cycle of treatment. Stringent complete response (sCR): Normal free light chain (FLC) ration, plus criteria for complete response. Complete response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in the bone marrow. Very Good Partial Response(VGPR): Positive immunofixation but negative electrophoresis; ≥90% reduction in serum M-component; Urine M-component ≤ 100mg per 24 hours. Partial Response (PR): ≥50% reduction in serum M-component and/or Urine M-component ≥90% reduction or < 200mg per 24 hours.

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events. | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Adverse Events (AE) are assessed according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 3.0. The maximum grade for each type of AE will be recorded for each patient. Grade 1: Mild AE. Grade 2: Moderate AE. Grade 3: Severe AE. Grade 4: Life-threatening or disabling AE. Grade 5: Death related AE.
Overall Survival (OS) | 2 years
  Survival time is defined as the time from registration to death due to any cause.
Progression Free Survival (PFS) | 2 years
  PFS is defined as the time from registration to the earliest date of documented disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death.
Duration of Response (DOR) | 2 years
  Duration of response will be calculated from the date of first evidence of response until the date of progression in the subset of patients with confirmed hematologic responses.

CONTACTS AND LOCATIONS:
Overall Officials: Jinxiang Fu, M.D., PhD, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China